CLINICAL TRIAL: NCT01615783
Title: Clinical and Economic Burden of Patients With Chronic Obstructive Pulmonary Disease in a Medicaid Population
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113900
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Costs; Resource utilization; Medicaid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medicaid beneficiaries: Medicaid beneficiaries with at least one medical or pharmacy claim during each year in the identification period (2004-2006)
  Interventions: Other: Subjects with COPD; Other: Subjects without COPD

INTERVENTIONS:
Other: Subjects with COPD — Medicaid beneficiaries diagnosed with Chronic Obstructive Pulmonary Disease (COPD) and newly initiated on a maintenance medication
Other: Subjects without COPD — Medicaid beneficiaries without a COPD diagnosis but having at least one medical or pharmacy claim during each year of the identification period

SUMMARY:
Reports suggest that the Medicaid population includes a higher percentage of smokers than the general population. A high prevalence of smokers in a population is likely to lead to a higher burden of chronic obstructive pulmonary disease (COPD). Few studies have evaluated the economic burden of COPD in a Medicaid population. The objective of this observational, retrospective cohort study is to estimate the economic burden of COPD in subjects with a COPD diagnosis who are enrolled in Medicaid and are receiving maintenance treatment covered by Medicaid.

Specifically, the null hypothesis for the primary outcome measure is that no difference is observed in all-cause costs between subjects with and without COPD. The test hypothesis is that there is a difference in all-cause costs between subjects with and without COPD.

Secondary outcomes to be evaluated include all-cause resource use and COPD-related costs for the COPD cohort.

The study uses a medical and pharmacy administrative claims database called MarketScan Medicaid Database that contains the medical, surgical, and prescription drug experience of nearly 7 million Medicaid recipients. This analysis will use data from 8 states.

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age at index date
* continuously eligible to receive healthcare services through Medicaid in the pre-index and follow-up period
* enrolled in fee-for-service plans
* without a diagnosis code of exclusionary comorbid conditions - cystic fibrosis, bronchiectasis, respiratory cancer, pulmonary fibrosis, pneumoconiosis, sarcoidosis, pulmonary tuberculosis (including fibrosis due to tuberculosis)

Exclusion Criteria:

* age less than 40 at index dates

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medicaid recipients (aged >=40 years) diagnosed with COPD (International Classification of Disease, Ninth Revision, Clinical Modification (ICD-9 CM) codes: 491.xx, 492.x, 496.xx) and newly initiated on Chronic Obstructive Pulmonary Disease (COPD) maintenance medication (maintenance therapies include ipratropium alone/combination ipratropium-albuterol (IPR), tiotropium (TIO), inhaled corticosteroid (ICS), long-acting beta-agonist (LABA), and combination product of inhaled corticosteroid and long-acting beta-agonist (ICS/LABA)) will be identified and matched in a 1 to 3 ratio to non-COPD Medicaid recipients on age (exact), gender, race, index year, Medicare dual eligibility, pre-index long-term care use. Index date was defined as the date of the first chronologically-occurring COPD maintenance medication during an identification period (01/01/2004 to 12/31/2006) for COPD patients, and as the date of the first medical or prescription claim during the index year of the corresponding matche
Sampling Method: Non-Probability Sample
Enrollment: 40884 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Incremental costs of COPD | 1 year
  Mean difference in all-cause costs between subjects with and without COPD. Incremental total costs and components of incremental total costs including pharmacy, medical, and long-term care will be reported

SECONDARY OUTCOMES:
All-cause resource use | 1 year
  The mean number of visits of each type of medical resource use including inpatient hospitalizations, emergency department [ED] visits, physician visits, outpatient visits, home healthcare visits/durable medical equipment, and long-term care visits.
COPD-related costs | 1 year
  Mean total, pharmacy, medical and long-term care costs associated with COPD in the cohort of subjects with a COPD diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline